CLINICAL TRIAL: NCT06749886
Title: An Exploratory Study of Tislelizumab in Combination with Chemotherapy in Immuno-experienced Patients with EGFR/ALK/ROS1-negative Advanced NSCLC in the Second-line Setting
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Chunxia Su, Director of the Clinical Research Center, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024LY0208
Record Dates: First submitted 2024-12-12; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Denosumab; tislelizumab; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- cohort1 (Experimental): The subjects in this cohort will receive denosumab combined with tislelizumab and docetaxel.
  Interventions: Drug: Denosumab; Drug: tislelizumab; Drug: Docetaxel

INTERVENTIONS:
Drug: Denosumab — Denosumab, 120 mg subcutaneous injection, every 21-28 days a cycle, given on the first day, a loading dose is given on d8 of the first cycle, and continued use
Drug: tislelizumab — Tislelizumab, 200 mg intravenous infusion, every 21 days a cycle, given on the first day, and continued use
Drug: Docetaxel — Docetaxel, 60 mg/m2 intravenous infusion, every 21 days a cycle, given on the first day, and continued use.

SUMMARY:
The goal of this clinical trial is to explore the efficacy and safety of denosumab in combination with tislelizumab and chemotherapy in the second-line treatment of immuno-experienced patients with EGFR/ALK/ROS1-negative advanced NSCLC.

Primary endpoint:

progression-free survival (PFS) assessed by investigators according to RECIST 1.1;

Secondary endpoint:

1. Overall survival (OS) assessed by investigators according to RECIST 1.1;
2. Objective response rate (ORR) assessed by investigators according to RECIST 1.1;
3. Disease control rate (DCR) assessed by investigators according to RECIST 1.1;
4. Duration of response (DOR) assessed by investigators according to RECIST 1.1;

Exploratory endpoint:

bone metastasis-free survival.

Participants will receive denosumab combined with tislelizumab and docetaxel.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥ 18 years old;
2. Patients with histologically or cytologically confirmed non-bone metastases stage IV NSCLC;
3. EGFR, ALK, and ROS1 are all wild-type (for other driver genes, if there is no first-line approval for corresponding targeted therapy or if the patient refuses targeted therapy, these patients are allowed to be enrolled);
4. first-line treatment with immune checkpoint inhibitors and clinical benefit (PFS ≥ 3 months);
5. Have measurable lesions (according to RECIST 1.1 criteria, the long diameter of CT scan of tumor lesions is ≥10mm, the short diameter of CT scan of lymph node lesions is ≥15mm, and the thickness of the scanning layer is not more than 5mm, and the measurable lesions have not received local treatment such as radiotherapy and cryotherapy);
6. ECOG PS: 0-2 points;
7. Estimated survival time≥ 3 months;
8. Adequate hematologic function, defined as absolute neutrophil count ≥1.5×109/L, platelet count ≥ 80×109/L, hemoglobin ≥ 90g/L (no history of blood transfusion within 7 days, not corrected with G-CSF and other hematopoietic stimulating factors);
9. adequate liver function, defined as total bilirubin levels ≤1.5 times the upper limit of normal (ULN) and aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels ≤ 2.5 times ULN, or for patients with liver metastases, AST and ALT levels ≤ 5 times ULN;
10. adequate renal function, defined as creatinine clearance ≥50ml/min (Cockcroft-Gault formula);
11. Adequate coagulation function, defined as the international normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 times ULN;
12. For female subjects of childbearing age, a negative urine or serum pregnancy test should be performed within 3 days prior to receiving the first dose of study drug, and if the urine pregnancy test result cannot be confirmed as negative, a blood pregnancy test is required;
13. If there is a risk of conception, male and female patients need to use highly effective contraception (i.e., a method with a failure rate of less than 1% per year) and continue until at least 180 days after stopping the trial treatment (Note: abstinence can be accepted as a contraceptive method if abstinence is the subject's usual lifestyle and preferred contraceptive method);
14. Subjects voluntarily joined this study, signed a written informed consent form before the implementation of any trial-related procedures, had good compliance, and cooperated with follow-up.

Exclusion Criteria:

1. Patients on first-line docetaxel chemotherapy;
2. Patients with symptomatic brain metastases (symptoms of brain metastases remain clinically stable for at least 1 month after treatment, and no steroids and anticonvulsants can be enrolled for at least 1 month before entering the study);
3. Presence of clinically uncontrollable pleural effusion/ascites effusion (patients who do not need to drain the effusion or who have stopped draining for 3 days without a significant increase in effusion can be enrolled);
4. have not recovered adequately from toxicity and/or complications caused by any intervention (i.e., ≤ grade 1 or to baseline, excluding fatigue or alopecia, prior to initiation of treatment);
5. Diagnosis of other malignant tumors within 5 years before the first dose, excluding radically treated basal cell carcinoma of the skin, squamous cell carcinoma of the skin and/or carcinoma in situ that has undergone radical resection, if other malignant tumors or lung cancer are diagnosed more than 5 years before administration, pathological or cytological diagnosis of recurrent metastatic lesions is required;
6. Active hemoptysis, active diverticulitis, intra-abdominal abscess, gastrointestinal obstruction and peritoneal metastasis requiring clinical intervention;
7. Received solid organ or blood system transplantation;
8. Class III-IV congestive heart failure (New York Heart Association classification), poorly controlled and clinically significant arrhythmia;
9. Active autoimmune disease requiring systemic treatment (such as the use of disease-modifying drugs, corticosteroids, or immunosuppressants) within 2 years prior to the first dose. Replacement therapies (e.g., thyroxine, insulin, or physiologic corticosteroids for adrenal or pituitary insufficiency) are not considered systemic therapy;
10. Patients who need long-term systemic use of corticosteroids (patients who need intermittent use of bronchodilators, inhaled corticosteroids, or local corticosteroids due to COPD and asthma can be enrolled);
11. History of non-infectious pneumonitis requiring corticosteroid treatment within 1 year before the first dose;
12. Have an active infection requiring treatment or have used systemic anti-infective drugs within one week before the first dose;
13. Known psychiatric illness or substance abuse that may affect compliance with trial requirements;
14. Those who are considered unsuitable for inclusion by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-11-19 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
progress free survival | up to 24 months
  Progression-free survival refers to the time from the start of combined treatment to any objectively documented tumor progression or patient death (the last follow-up date for patients lost to follow-up; the end of follow-up date for patients still alive at the end of the study).

SECONDARY OUTCOMES:
overall survival | up to 24 months
  Overall survival (OS): the time from the first dose to death from any cause (the last follow-up date for patients who were lost to follow-up; the end of follow-up date for patients who were still alive at the end of the study)
objective response rate | 12 months
  Objective response rate (ORR) refers to the proportion of patients whose tumors shrink to a certain amount and remain so for a certain period of time, including cases of complete remission (CR) and partial remission (PR).
Disease control rate | 12 months
  Disease control rate (DCR): refers to the proportion of patients whose tumors shrink to a certain amount and remain so for a certain period of time, including cases of complete remission (CR), partial remission (PR) and stable disease (SD).
Duration of remission | 12 months
  Duration of response (DOR): refers to the duration from the first recorded confirmed response (CR or PR) to the first recorded disease progression (PD) or death due to any cause (whichever occurs first).

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No